CLINICAL TRIAL: NCT01552005
Title: Description of Drug Utilization and Assessment of Impact of Saxagliptin on Health Status of Patients With Type 2 Diabetes in France
Acronym: DIAPAZON
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: CV181-148
Record Dates: First submitted 2012-02-09; First posted 2012-03-13 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Type 2 Diabetes Mellitus (T2D)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Population of patients treated with Saxagliptin
  Interventions: Drug: Saxagliptin

INTERVENTIONS:
Drug: Saxagliptin — No Intervention

SUMMARY:
The purpose of this study is to respond to The French Health Authority which has requested BMS France and Astra Zeneca (AZ) France to set-up a long-term cohort study in a representative sample of French Type 2 Diabetes mellitus (T2D) patients treated with Saxagliptin to generate real world data on drug utilization, joint population, non comparative effectiveness and safety

DETAILED DESCRIPTION:
Time Perspective: Ambispective cohort follow by a 18 to 24 month follow up period, Retrospective follow by Prospective.

ELIGIBILITY:
Inclusion Criteria:

* Registry

  * Patient ≥ 18 years old
  * Patient with T2D
* Ambispective Cohort

  * Patient ≥ 18 years old
  * Patient with T2D
  * Patient initiated with Saxagliptin in the last 6 months before the inclusion or day of inclusion visit (whatever his/her ongoing hypoglycaemic treatment)
  * Patient agreeing to participate, and not yet enrolled by another physician

Exclusion Criteria:

* Patient participating in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be proposed by GPs and diabetologists in France to ambulatory patients
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Evolution of Glycated hemoglobin (HbA1c) level, weight and the onset of hypoglycemic over time (2 years) for patients treated with Saxagliptin | 24 months
  HbA1c level <7% at Y2, weight and assessment of hypoglycaemic events after a 2-year exposure to Saxagliptin
Joint population of Saxagliptin based on socio-demographic data, medical history, disease history, comorbidities including renal, hepatic and cardiac functions, HbA1c level at treatment initiation) | One year (average)
Utilization of Saxagliptin by General practitioners (GPs) and diabetologists in France (based on indication, initial dosage and adjustments, co-prescriptions, glycemic monitoring) | During the treatment (Up to 2 years)
Retention rate of Saxagliptin and to describe discontinuation rate and reasons | At 2 years

SECONDARY OUTCOMES:
Distribution of different hypoglycaemic therapeutic strategies used in France and characteristics of T2D patients depending on therapeutic strategies | 2 month
Saxagliptin utilization according to patient's profile and disease characteristics | 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3663&filename=CSR_D1680R00018_CV181_148.pdf